CLINICAL TRIAL: NCT00693459
Title: Feasibility Study of a New Circular Anal Dilator for Transanal Hemorrhoidectomy
Brief Title: Study of a New Circular Anal Dilator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 07-07-06
Record Dates: First submitted 2008-02-27; First posted 2008-06-09 (Estimated); Last update posted 2022-08-15 (Actual); Status verified 2013-01

CONDITIONS: Hemorrhoids
Keywords: Hemorrhoids
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Circular anal dilator (Other): Circular anal dilator group-An anoscope has been developed that outlines the precise path for hemorrhoid excision. This instrument allows a modified Ferguson hemorrhoidectomy to be performed and does not alter the steps of the operation.
  Interventions: Device: Circular Anal Dilator for Transanal Hemorrhoidectomy

INTERVENTIONS:
Device: Circular Anal Dilator for Transanal Hemorrhoidectomy — The Circular Anal Dilator for Transanal Hemorrhoidectomy (product #CAD01) allows the standard of care Ferguson hemorrhoidectomy to be performed and does not alter the steps of the operation. The presumed advantages are the ability of the dilator to guide an accurate dissection and also to decrease the overall time it takes to perform hemorrhoidectomy.
  Other Names: Chemo 2

SUMMARY:
The purpose of this research study is to test the effectiveness of a new anoscope used while performing a traditional hemorrhoidectomy.

DETAILED DESCRIPTION:
Historically, surgical hemorrhoidectomy has been effective at eliminating hemorrhoids but is associated with high complication rates and post-operative disability. The problems that are most common immediately after hemorrhoidectomy are severe pain, urinary retention, bleeding and fecal impaction. The most dreaded long term complications are anal stricture and fecal incontinence.

Stricture or narrowing of the anal canal after hemorrhoidectomy is the direct result of excising too much anoderm and mucosa. Even in circumferential prolapsed hemorrhoids, a standard three quadrant hemorrhoidectomy is all that is necessary. Mild anal stricture can be treated with a Hegar dilator but severe stricture requires a lateral internal sphincterotomy with or without a skin advancement flap. These operations are morbid and results are generally poor.

Anal sensation is partially impaired leading to some degree of incontinence of 50% of patients after hemorrhoidectomy. Persistent incontinence results from being over aggressive during the hemorrhoidectomy and excising muscle with the hemorrhoid during dissection.

The majority of these long term complications are solely dependent on surgical technique. The majority of hemorrhoidectomies performed today are still performed by non-specialty surgeons. They rely on various instruments during the surgery to perform the operation in the anal canal with adequate exposure but the most important instrument is the anoscope.

A variety of anoscopes are currently available, but the standard anoscope used for hemorrhoidectomy is the Hill-Ferguson. The Hill-Ferguson is a crescent shaped instrument that provides adequate exposure in the anal canal and allows the surgeon to perform a Ferguson hemorrhoidectomy, the standard of care for hemorrhoidectomy in this country. During this procedure an elliptical excision is begun at the perianal skin to include both external and internal hemorrhoids and is ended at the anorectal ring. A full thickness of mucosa and submucosa is excised and the surgeon should dissect superficial to the internal sphincter muscle. The strip of this excision should be no wider than 1.5 cm but currently nothing prevents the surgeon from exceeding this limitation or from taking muscle with the excision. The widely accepted Hill-Ferguson Anoscopes provide vast exposure but do not set any boundaries for the surgeon when performing this operation.

Over the last several decades few modifications have been introduced to alter the contour of the anoscope in an attempt to reduce the complications of post-operative stricture and incontinence. Furthermore, the current anoscopes lack the ability to outline a precise excision path for the infrequent anorectal surgeon or for the non-specialist in the community.

Recently, Ethicon surgical has developed an anoscope that outlines the precise path for hemorrhoid excision without the possibility of excision greater than 1.5 cm of anoderm with each excision. This instrument allows the standard of care Ferguson hemorrhoidectomy to be performed and does not alter the steps of the operation. The presumed advantages are the ability of the instrument to guide an accurate dissection and also to decrease the overall time it takes to perform hemorrhoidectomy. It has been tested in several porcine models. Operative times, tissue excised, and evaluation of the suture line were addressed during these trials and there were no instances of bleeding or excessive tissue excision.

The study design will be a prospective feasibility trial. Patients who are scheduled for operative excisional hemorrhoidectomy will undergo their planned procedure according to the standard of care which is a Ferguson hemorrhoidectomy. The only new variable introduced will be the application of a new anoscope to facilitate the dissection. Other than the new anoscope all pre-operative, intra-operative, and post-operative guidelines consistent with the current standards will be followed. The primary goal is to confirm that the new anoscope permits standard hemorrhoidectomy, and to obtain phase I data confirming that this novel anoscope is safe and efficacious in the performance of a Ferguson hemorrhoidectomy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with internal or external symptomatic hemorrhoids.
* Subjects who have failed, or are not suitable for office management of their hemorrhoids.
* Subjects who are 18 years of age and older
* Subjects of either gender
* Subjects, who are willing and able to adhere to protocol requirements, agree to participate in the study program and provide written and informed consent

Exclusion Criteria:

* Subjects who have had previous hemorrhoid surgery.
* Subjects with internal hemorrhoids that may be suitable for office management.
* Subjects with incontinence.
* Subjects with evidence of acute sepsis or the presence of a fistula.
* Subjects with a medical condition that may interfere with the evaluation of safety or effectiveness of the study device.
* Subjects who have another condition that in the opinion of the investigator precludes further participation in the study.
* Subjects with an anal stricture.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of the new device by the number of participants with Adverse Events | 1 year post-operative
  This study will be monitored to ensure the identification, documentation and analysis of all adverse events in regards to safety and efficacy of the new device. All adverse events, unforeseen or otherwise will be recorded as data. Information will be reported on the 1)Visual Analog Pain scores, 2)Incontinence score, using the Wexner Oliveira score, 3) Presence of Stenosis 4) Continued bleeding or symptoms, 5) Wound Infection, 6) Bladder Retention

SECONDARY OUTCOMES:
Evaluate the efficacy of the new device by the number of participants with Adverse Events | 1 year post operative
  This study will be monitored to ensure the identification, documentation and analysis of all adverse events in regards to safety and efficacy of the new device. All adverse events, unforeseen or otherwise will be recorded as data. Information will be reported on the 1)Visual Analog Pain scores, 2)Incontinence score, using the Wexner Oliveira score, 3) Presence of Stenosis 4) Continued bleeding or symptoms, 5) Wound Infection, 6) Bladder Retention

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Champagne, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals of Cleveland Case Medical Center, Cleveland, Ohio, United States